CLINICAL TRIAL: NCT04676945
Title: Analysis of Risk in MDS Over Time - Comparison of Treated vs Untreated Patients
Status: Completed | Type: Observational
Sponsor: Michael Pfeilstöcker (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor-Investigator, Michael Pfeilstöcker, Univ.Prof.Dr.med.univ., Mein Hanusch-Krankenhaus
Organization: Mein Hanusch-Krankenhaus (Other)
Other Study IDs: N/A-NI-MDSAML-PI-14023
Record Dates: First submitted 2020-11-26; First posted 2020-12-21 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Myelodysplastic Syndromes
Keywords: MDS; IPSS-R
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- untreated control group: NO MDS disease modifying therapy
- treated patients: ANY MDS disease modifying therapy

SUMMARY:
A comparison of treated vs untreated patients with MDS with a sample size of approximately 8000 patients in 11 countries.

DETAILED DESCRIPTION:
Non-interventional multicentre retrospective study using chart reviews - study was submitted to the ethics committee of city of Vienna - due to the design of the study no specific approval necessary.

Inclusion of MDS (all subtypes and risk groups) patients according to WHO or oligoblastic AML (RAEB-T according to FAB), untreated and treated during their chronic MDS phase

The 26 centers of the IWG-PM have provided control data set of untreated, all centers will be asked for contribution of treated patients Data will be collected in Austria, Brazil, Czech Republic, France, Germany, Italy, Japan, Netherlands, Spain, UK, USA.

ELIGIBILITY:
Inclusion Criteria:

* MDS (all subtypes and risk groups) according to WHO or oligoblastic AML (RAEB-T according to FAB) patients untreated and treated during their chronic MDS phase

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: MDS (all subtypes and risk groups) according to WHO or oligoblastic AML (RAEB-T according to FAB) patients untreated and treated during their chronic MDS phase Population derived from registries of participating centres.
Sampling Method: Non-Probability Sample
Enrollment: 9179 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2022-11-21 (Actual)

PRIMARY OUTCOMES:
1.Overall Survival | From date of diagnosis until the date of death or lost to follow-up, whichever came first. No administrative censoring will be applied to the retrospectively collected data, a minimum period of two months of stable disease will be required.
  In *overall survival* two possible events are defined:
  * *death* (regarded as complete observation)
  * *end of follow up* (regarded as censored observation) Time is calculated from diagnosis to the first occurrence of one of the above listed events.
2.Time to transformation | From date of diagnosis until the date of transformation,death or lost to follow-up, whichever came first. No administrative censoring will be applied to the retrospectively collected data,a minimum period of two months of stable disease will be required.
  In *time to transformation* three possible events are defined:
  * *transformation into AML* (regarded as complete observation)
  * *death without transformation* (regarded as censored observation)
  * *end of follow up* (regarded as censored observation) Time is calculated from diagnosis to the first occurrence of one of the above listed events.
  In case of *transformation into AML* this results in a complete observation, in case of *death without transformation* or *end of follow up* the observation is treated as censored.

CONTACTS AND LOCATIONS:
Locations (1):
- Hanusch Krankenhaus, 3.Medizinische Abteilung, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Greenberg PL, Tuechler H, Schanz J, Sanz G, Garcia-Manero G, Sole F, Bennett JM, Bowen D, Fenaux P, Dreyfus F, Kantarjian H, Kuendgen A, Levis A, Malcovati L, Cazzola M, Cermak J, Fonatsch C, Le Beau MM, Slovak ML, Krieger O, Luebbert M, Maciejewski J, Magalhaes SM, Miyazaki Y, Pfeilstocker M, Sekeres M, Sperr WR, Stauder R, Tauro S, Valent P, Vallespi T, van de Loosdrecht AA, Germing U, Haase D. Revised international prognostic scoring system for myelodysplastic syndromes. Blood. 2012 Sep 20;120(12):2454-65. doi: 10.1182/blood-2012-03-420489. Epub 2012 Jun 27. PMID 22740453
- [Background] Lamarque M, Raynaud S, Itzykson R, Thepot S, Quesnel B, Dreyfus F, Rauzy OB, Turlure P, Vey N, Recher C, Dartigeas C, Legros L, Delaunay J, Visanica S, Stamatoullas A, Fenaux P, Ades L. The revised IPSS is a powerful tool to evaluate the outcome of MDS patients treated with azacitidine: the GFM experience. Blood. 2012 Dec 13;120(25):5084-5. doi: 10.1182/blood-2012-09-453555. No abstract available. PMID 23243156
- [Background] Montalban-Bravo G, Garcia-Manero G. Myelodysplastic syndromes: 2018 update on diagnosis, risk-stratification and management. Am J Hematol. 2018 Jan;93(1):129-147. doi: 10.1002/ajh.24930. PMID 29214694
- [Background] Sekeres MA, Swern AS, Fenaux P, Greenberg PL, Sanz GF, Bennett JM, Dreyfus F, List AF, Li JS, Sugrue MM. Validation of the IPSS-R in lenalidomide-treated, lower-risk myelodysplastic syndrome patients with del(5q). Blood Cancer J. 2014 Aug 29;4(8):e242. doi: 10.1038/bcj.2014.62. No abstract available. PMID 25171203
- [Background] Della Porta MG, Alessandrino EP, Bacigalupo A, van Lint MT, Malcovati L, Pascutto C, Falda M, Bernardi M, Onida F, Guidi S, Iori AP, Cerretti R, Marenco P, Pioltelli P, Angelucci E, Oneto R, Ripamonti F, Bernasconi P, Bosi A, Cazzola M, Rambaldi A; Gruppo Italiano Trapianto di Midollo Osseo. Predictive factors for the outcome of allogeneic transplantation in patients with MDS stratified according to the revised IPSS-R. Blood. 2014 Apr 10;123(15):2333-42. doi: 10.1182/blood-2013-12-542720. Epub 2014 Feb 20. PMID 24558201
- [Background] Pfeilstocker M, Tuchler H, Schonmetzler A, Nosslinger T, Pittermann E. Time changes in predictive power of established and recently proposed clinical, cytogenetical and comorbidity scores for Myelodysplastic Syndromes. Leuk Res. 2012 Feb;36(2):132-9. doi: 10.1016/j.leukres.2011.09.007. Epub 2011 Oct 2. PMID 21967831
- [Background] Pfeilstocker M, Tuechler H, Sanz G, Schanz J, Garcia-Manero G, Sole F, Bennett JM, Bowen D, Fenaux P, Dreyfus F, Kantarjian H, Kuendgen A, Malcovati L, Cazzola M, Cermak J, Fonatsch C, Le Beau MM, Slovak ML, Levis A, Luebbert M, Maciejewski J, Machherndl-Spandl S, Magalhaes SM, Miyazaki Y, Sekeres MA, Sperr WR, Stauder R, Tauro S, Valent P, Vallespi T, van de Loosdrecht AA, Germing U, Haase D, Greenberg PL. Time-dependent changes in mortality and transformation risk in MDS. Blood. 2016 Aug 18;128(7):902-10. doi: 10.1182/blood-2016-02-700054. Epub 2016 Jun 22. PMID 27335276